CLINICAL TRIAL: NCT02802592
Title: EPOgen and Restrictive Transfusions in Patients Undergoing Cardiac Surgery (EPORT)
Acronym: EPORT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00050961
Record Dates: First submitted 2016-06-03; First posted 2016-06-16 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Cardiac Surgery-CABG; Cardiac Valve Replacement
MeSH Terms: interventions — Epoetin Alfa; Erythropoietin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epogen (Active Comparator): 1000 IU/kg Epogen in 250 ml of normal saline infused over 1 hr
  Interventions: Drug: Epogen
- Normal Saline (Placebo Comparator): 250 ml normal saline infused over 1 hr
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Epogen — 1:1 randomization to either the Epogen arm or Placebo(Normal Saline) arm
  Other Names: EPOETIN; Procrit
  Arms: Epogen
Drug: Normal Saline — 1:1 randomization to either the Epogen arm or Placebo(Normal Saline) arm
  Other Names: Placebo
  Arms: Normal Saline

SUMMARY:
EPOgen and Restrictive Transfusions in Patients Undergoing Cardiac Surgery (EPORT)

DETAILED DESCRIPTION:
The investigator proposes a study investigating the use of restrictive transfusion triggers and administration of single preoperative high dose shot of epoetin alfa (rhEPO) in a young (age < 65 years of age) population undergoing cardiac surgery. The investigator believes that participants can tolerate a lower Hemoglobin (Hgb). Therefore, the control group will benefit from a restrictive transfusion trigger and experimental group will benefit from EPO providing a synergistic stimulus for erythropoiesis. This proposed study has potential to reduce overall transfusion utilization in cardiac surgery and improve standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female and 18 years of age or older, but less than 65 years of age
* Be willing to performed written informed consent prior to study initiation
* Be willing and able to comply with the protocol for study duration
* Be scheduled to undergo elective cardiac surgery requiring CPB and including: coronary artery bypass graft (CABG), aortic, mitral, or tricuspid valve replacement or repair, replacement of more than one cardiac valve, or CABG with combined cardiac valve replacement or repair.

Exclusion Criteria:

* Over the age of 64 years
* Patients who receive allogeneic transfusion 60 days prior to surgery
* Hgb > 15g/dl
* Patients who are pregnant or currently lactating
* Women of childbearing potential (e.g. those not surgically sterilized or not post-menopausal) must use 2 methods of contraception including at least one barrier method.
* End-stage renal disease requiring renal replacement therapy or dialysis
* Hepatic dysfunction (defined as total bilirubin value > 1.5 mg/dl)
* Off-pump (no CPB) cardiac surgery
* Emergency surgical procedure
* Inability to receive blood products
* Endocarditis as defined my Modified Duke Criteria
* Any congenital coagulation disorder
* Chronic anemia (defined as preoperative Hgb concentration < 10 g/dl)
* Low platelet count (defined as preoperative platelet count less than 150 x 103/μl)
* Not a surgical candidate due to high risk of morbidity or mortality
* Surgery for aneurysm repair, dissection, or other thoracic aortic procedure
* Congenital heart surgery
* Cardiogenic shock or hemodynamic instability within 24 hours prior to surgery, as defined by systolic blood pressure < 80 mmHg and heart rate > 120 beats per minute
* Known malignancy within the past 5 years
* Life expectancy < 12 months
* Current active infection requiring antibiotic treatment
* Inability to comply with study protocol
* Contraindication to Epogen
* Hypersensitivity to epoetin or any component of the formulation
* Pure red cell aplasia (due to epoetin or other epoetin protein drugs)
* Contraindication to Ferrous Sulfate
* Hypersensitivity to iron salts or any component of the formulation
* Hemochromatosis
* Hemolytic anemia
* In the opinion of the Principle Investigator (PI) any specific disease process or confounding variables that may inappropriately alter the outcome of the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06-15 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith A. Horvath, MD, Principal Investigator — Johns Hopkins Community Physicians
Locations (1):
- Suburban Hospital, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated due to loss of funding and those participants enrolled were not un-blinded to the study team members.
Groups:
- All Participants: 1000 IU/kg Epogen in 250 ml of normal saline infused over 1 hr Epogen: 1:1 randomization to either the Epogen arm or Placebo(Normal Saline) arm
  OR
  250 ml normal saline infused over 1 hr Normal Saline: 1:1 randomization to either the Epogen arm or Placebo(Normal Saline) arm
Period: Overall Study
Arm/Group | All Participants
Started | 4
Completed | 0
Not Completed | 4
Not completed — Study terminated due to loss of funding | 4

BASELINE CHARACTERISTICS:
Population: This study was terminated due to loss of funding and those participants enrolled were not un-blinded to the study team members.
Arm/Group | All Participants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Packed Red Blood Cells Transfused During the Intraoperative and Immediate Postoperative Period
Time Frame: Start of surgery to 96 hours post op
Population: This study was terminated prematurely due to a loss of funding. There is no data available for this outcome measure.
Arm/Group | Epogen | Normal Saline
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Length of Stay (# of Total Days Hospitalized)
Time Frame: up to one year from date of surgery
Population: This study was terminated prematurely due to a loss of funding. There is no data available for this outcome measure.
Arm/Group | Epogen | Normal Saline
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Hospitalization Cost
Time Frame: up to one year from date of surgery
Population: This study was terminated prematurely due to a loss of funding. There is no data available for this outcome measure.
Arm/Group | Epogen | Normal Saline
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Quality of Life as Assessed by Short Form-36 Quality of Life Survey
Time Frame: assessed at 1-week, 1-month, and 3-months from date of surgery
Population: This study was terminated prematurely due to a loss of funding. There is no data available for this outcome measure.
Arm/Group | Epogen | Normal Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=4)
Cerebrovascular Accident (Blood and lymphatic system disorders) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=4)
Mediastinal bleeding (Blood and lymphatic system disorders) | 1 (1)
Complete Heart Block (Cardiac disorders) | 1 (1)
Pleural Effusion (Blood and lymphatic system disorders) | 1 (1)
Acute Congestive Heart Failure (Cardiac disorders) | 1 (1)
Ankle Edema (Bilateral) (Blood and lymphatic system disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes